CLINICAL TRIAL: NCT05109871
Title: A Prospective Cross-sectional Study to Determine the Reliability and Validity of Inline 'Pull' Dynamometry for Measuring Peak Knee Extensor Torque in Patients Following Anterior Cruciate Ligament (ACL) Reconstruction: HRA & HCRW Approval Issued.
Brief Title: Reliability and Validity of Inline Dynamometry Study for Measuring Knee Extensor Torque
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SP0558
Record Dates: First submitted 2021-09-21; First posted 2021-11-05 (Actual); Results first posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2022-05

CONDITIONS: Anterior Cruciate Ligament Injuries; Anterior Cruciate Ligament Rupture; Anterior Cruciate Ligament Tear
Keywords: Dynamometer; Dynamometry; Hand held; Inline; Traction; Pull; Validity; Reliability
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Kforce Link (Experimental)
  Interventions: Other: KForce Link

INTERVENTIONS:
Other: KForce Link — Traction (pull-type) dynamometer

SUMMARY:
This study will investigate the reliability and validity of an inline 'pull-type' dynamometer for measuring peak knee extensor torque. For the reliability study, healthy volunteers will be assessed by two assessors (inter-rater) at the index testing session, with testing repeated by one assessor one week later (test-retest). Validity will be investigated against isometric electromechanical dynamometry (gold standard) in patients following anterior cruciate ligament (ACL) reconstruction.

DETAILED DESCRIPTION:
This is a prospective, cross sectional study using a within-participant, repeated measures design. The inter-rater and test-retest reliability of the KForce Link (pull-type dynamometer) will be determine using 50 healthy subjects. The validity of the KForce Link will be determined using 52 post-operative ACL reconstruction patients against the gold standard of isometric electromechanical dynamometry (Cybex). All testing will be performed isometrically with the knee positioned at 60 degrees knee flexion. Assessors and participants will be blinded to the scores until testing is complete.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* No contraindications to maximal force testing (see exclusion criteria).
* For the ACL reconstruction participant cohort: diagnosed with ACL injury that was managed with ACL reconstruction surgery, with or without additional meniscal surgery. If medicated, stable dose of current regular medication for at least 4 weeks prior to study entry.
* For the healthy control participant cohort: no current or previous history of significant lower limb injury, or a history of previous minor injury that is symptomatic at the time of recruitment. No previous lower limb surgery. No course of medication, whether prescribed or over the counter, other than vitamins and mineral supplements or, for females, oral contraceptives.

Exclusion Criteria:

* Unable to provide written consent to study participation, or there are contraindications to maximal force testing, including the following:

  * History of chronic disease or disorder that may put the participants at risk because of participation in the study including non-united fractures, epilepsy, cardiac insufficiency, severe peripheral vascular disease, aneurysms, anticoagulant therapy, recent (<3 months) radiotherapy or chemotherapy, long term steroid use (>3 months), pregnancy, neurological disorders (e.g., Parkinson's disease), skin conditions at point of force testing, severe osteoporosis, malignancy, rheumatoid arthritis.
* Conditions or symptoms that may influence the result of the study, or the participant's ability to participate in the study including pain, limited range of motion, knee effusion, or anaemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Norris, BSc, Principal Investigator — Aintree University Hospital
Locations (1):
- Aintree University Hospital, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stark T, Walker B, Phillips JK, Fejer R, Beck R. Hand-held dynamometry correlation with the gold standard isokinetic dynamometry: a systematic review. PM R. 2011 May;3(5):472-9. doi: 10.1016/j.pmrj.2010.10.025. PMID 21570036
- [Background] Whiteley R, Jacobsen P, Prior S, Skazalski C, Otten R, Johnson A. Correlation of isokinetic and novel hand-held dynamometry measures of knee flexion and extension strength testing. J Sci Med Sport. 2012 Sep;15(5):444-50. doi: 10.1016/j.jsams.2012.01.003. Epub 2012 Mar 15. PMID 22424705
- [Background] Bohannon RW, Bubela DJ, Wang YC, Magasi SR, Gershon RC. Adequacy of belt-stabilized testing of knee extension strength. J Strength Cond Res. 2011 Jul;25(7):1963-7. doi: 10.1519/JSC.0b013e3181e4f5ce. PMID 21399535
- [Background] Kelln BM, McKeon PO, Gontkof LM, Hertel J. Hand-held dynamometry: reliability of lower extremity muscle testing in healthy, physically active,young adults. J Sport Rehabil. 2008 May;17(2):160-70. doi: 10.1123/jsr.17.2.160. PMID 18515915
- [Background] Hansen EM, McCartney CN, Sweeney RS, Palimenio MR, Grindstaff TL. Hand-held Dynamometer Positioning Impacts Discomfort During Quadriceps Strength Testing: A Validity and Reliability Study. Int J Sports Phys Ther. 2015 Feb;10(1):62-8. PMID 25709864
- [Background] Sinacore JA, Evans AM, Lynch BN, Joreitz RE, Irrgang JJ, Lynch AD. Diagnostic Accuracy of Handheld Dynamometry and 1-Repetition-Maximum Tests for Identifying Meaningful Quadriceps Strength Asymmetries. J Orthop Sports Phys Ther. 2017 Feb;47(2):97-107. doi: 10.2519/jospt.2017.6651. PMID 28142362
- [Background] Almeida GPL, Albano TR, Melo AKP. Hand-held dynamometer identifies asymmetries in torque of the quadriceps muscle after anterior cruciate ligament reconstruction. Knee Surg Sports Traumatol Arthrosc. 2019 Aug;27(8):2494-2501. doi: 10.1007/s00167-018-5245-3. Epub 2018 Oct 30. PMID 30377716
- [Background] Suzuki T. Reliability of measurements of knee extensor muscle strength using a pull-type hand-held dynamometer. J Phys Ther Sci. 2015 Mar;27(3):967-71. doi: 10.1589/jpts.27.967. Epub 2015 Mar 31. PMID 25931771
- [Derived] Norris R, Morrison S, Price A, Pulford S, Meira E, O'Neill S, Williams H, Maddox TW, Carter P, Oldershaw RA. Inline dynamometry provides reliable measurements of quadriceps strength in healthy and ACL-reconstructed individuals and is a valid substitute for isometric electromechanical dynamometry following ACL reconstruction. Knee. 2024 Jan;46:136-147. doi: 10.1016/j.knee.2023.12.006. Epub 2023 Dec 23. PMID 38142660

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For inter- and intra-rater reliability of ID in a healthy cohort, 52 participants was recruited from Liverpool University Hospitals, NHS Foundation Trust (LUHFT). For intra-rater reliability and criterion validity in an ACL-reconstructed cohort, consecutive patients presenting to an orthopaedic outpatient clinic following ACL reconstruction, were recruited from LUHFT. Testing sessions were conducted in a LUHFT physiotherapy department between September 2021 and August 2022.
Groups:
- Healthy Participants: Fifty healthy participants tested to determine the inter- and intra-rater reliability of inline dynamometry
- ACL Reconstructed Participants: For intra-rater reliability and criterion validity in an ACL-reconstructed cohort, 52 consecutive patients presenting to an orthopaedic outpatient clinic following ACL reconstruction, with or without concomitant meniscal repair or excision, were recruited from LUHFT.
Period: Overall Study
Arm/Group | Healthy Participants | ACL Reconstructed Participants
Started | 50 | 52
Completed | 50 | 52
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 102 (50 healthy, 52 ACL-reconstructed)
Groups:
- Healthy Participants: Fifty participants (25 females and 25 males) were recruited to determine the inter- and intra-rater reliability of ID in a healthy cohort
- ACL-reconstructed Participants: Fifty two participants (5 females and 47 males) were recruited to determine the intra-rater reliability and validity of ID in an ACL-reconstructed cohort.
- Total: Total of all reporting groups
Arm/Group | Healthy Participants | ACL-reconstructed Participants | Total
Number analyzed (Participants) | 50 | 52 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 52 | 102
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 5 | 30
  Male | 25 | 47 | 72
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 47 | 49 | 96
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 50 | 52 | 102

OUTCOME MEASURES:

1. Primary Outcome: Peak Knee Extensor Torque Measured in Newton Metres Per kg (Nm/kg)
Description: Peak knee extensor force (N) multiplied by lever length (m), normalised to body weight (kg)
Time Frame: 30 minutes
Measure: Mean (Standard Deviation); unit: Newton metres per kg
Groups:
- ACL Reconstructed Participants: For intra-rater reliability and criterion validity in an ACL-reconstructed cohort, 56 consecutive patients presenting to an orthopaedic outpatient clinic following ACL reconstruction, with or without concomitant meniscal repair or excision, were recruited from LUHFT.
Arm/Group | Healthy Participants | ACL Reconstructed Participants
Number analyzed (Participants) | 50 | 52
Newton metres per kg | 3.12 (0.66) | 2.66 (0.66)

2. Secondary Outcome: Pain During Testing on a Numerical Rating Scale (0-10)
Description: Numerical rating scale of pain from 0 to 10, with 0 indicating no pain (better outcome) and 10 indicating worst pain possible (worse outcome).
Time Frame: 45 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Healthy Participants | ACL Reconstructed Participants
Number analyzed (Participants) | 50 | 52
score on a scale | 1 [0 to 2] | 1 [0 to 3]

ADVERSE EVENTS:
Time Frame: Through study completion, on average 12 weeks
Description: As per Clinical trials descriptions
Arm/Group | Healthy Participants | ACL Reconstructed Participants
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/52
Other Adverse Events (participants affected / at risk) | 0/50 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-19): https://cdn.clinicaltrials.gov/large-docs/71/NCT05109871/Prot_SAP_000.pdf